CLINICAL TRIAL: NCT01187446
Title: A Multicenter, Open-label, Randomized, Phase I/II Study Evaluating the Safety and Efficacy of Low-dose (12 Gy) Total Skin Electron Beam Therapy (TSEBT) Combined With Vorinostat Versus Low-dose TSEBT Monotherapy in Mycosis Fungoides (MF)
Brief Title: Low-dose (12 Gy) TSEBT+Vorinostat Versus Low-dose TSEBT Monotherapy in Mycosis Fungoides
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision by funding source
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Youn Kim, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18417; SU-08092010-6685 (Other: Stanford University); LYMNHL0078 (Other: OnCore)
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Cutaneous Lymphoma; Cutaneous T-cell Lymphoma
Keywords: Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TSEBT & Vorinostat (Experimental): Total skin electron beam therapy (TSEBT) will be performed per institution guidelines.
  Vorinostat will be administered at a dose of 400 mg/day, starting one day prior to the initiation of TSEBT. During TSEBT, vorinostat should be taken in the morning and preferably prior to TSEBT.
  Interventions: Radiation: Total skin electron beam therapy (TSEBT); Drug: Vorinostat
- TSEBT only (Active Comparator): Total skin electron beam therapy (TSEBT) will be administered according to the Stanford 6-field technique or equivalent technique per institutional standards. Patients will receive a planned total skin dose of 12 grey (Gy) fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment); 4 days each week; for a total of 3 weeks. Supplements will routinely be applied to the perineum and soles as well as any other "shadowed" sites involved by disease, such as the inframammary regions (1-2 Gy fractions to a total dose of 12 Gy). Discrete tumors may receive additional "boost" treatment not to exceed 12 Gy.
  Interventions: Radiation: Total skin electron beam therapy (TSEBT)

INTERVENTIONS:
Radiation: Total skin electron beam therapy (TSEBT) — TSEBT is administered as 12 Gy fractionated at 2 grey (Gy)/cycle (each cycle requiring 2 days of treatment); 4 days each week; for 3 weeks.
Drug: Vorinostat — Starting doses of is vorinostat 400 mg/day, continuing for 8 weeks.
  Other Names: Zolinza
  Arms: TSEBT & Vorinostat

SUMMARY:
The purpose of this study is to determine if vorinostat combined with low-dose total skin electron beam therapy (TSEBT) offers superior clinical benefit (efficacy & safety) over low-dose TSEBT alone in participants with mycosis fungoides (MF)

Treatment in this study is TSEBT +/- vorinostat, with participants stratified by MF stage.

DETAILED DESCRIPTION:
Vorinostat is a histone deacetylase inhibitor (HDAC) that is FDA-approved for treatment of mycosis fungoides (MF), and has shown activity as a radiation-sensitizer in preclinical studies. Treatment of various cell lines [glioblastoma multiforme (GBM), non-small cell lung cancer (NSCLC), melanoma] has shown that pretreatment with vorinostat had a significant effect on radiation kill. This effect is believed to be secondary to multiple mechanisms that may involve antiproliferative growth inhibition and effects on DNA repair after exposure to radiation. A histone deacetylase inhibitor such as vorinostat may act as a radiosensitizer by modulating the expression of single- and double-strand DNA repair proteins such as KU67, KU86, H2AX, and Rad50. These DNA repair proteins are enzymes of that repair radiation-induced damage. The decrease in these DNA repair enzymes is thought to be the key mechanism of sensitization. Down-regulation of several key proteins involved in the nonhomologous end joining pathway is thought to generate a G2/M checkpoint blockade. Vorinostat may also cause an "open chromatin" structure increasing the effect of radiation damage to DNA. This is exemplified by the finding that there is a prolonged H2AX phosphorylation and H2AX foci formation. The mechanism producing this prolongation of H2AX foci is thought to contribute to the damage, and thus killing effect of the radiation.

In the pivotal phase 2 trial of vorinostat, an overall response rate of nearly 30% was reported. The median time to progression was 4.9 months overall, and 9.8 months for MF stage IIB or higher responders. Through hyperacetylation of both histone and non-histone proteins, vorinostat is felt to exert its anti-tumor activity via several mechanisms, including cell cycle arrest, induction of apoptosis, reactive oxygen species generation, cell differentiation, and angiogenesis inhibition. Importantly, a number of pre-clinical studies have reported on the potential of vorinostat to enhance radiosensitivity of several different human tumor cell lines. The rational for clinical trial investigating combination of vorinostat and TSEBT not only comes from their underlying mechanism for potential synergy as suggested by prior in-vitro studies but also due to general therapeutic advantage derived from their non-overlapping toxicities.

Recent results from a phase 1 dose-escalation trial combining palliative pelvic radiation (30 Gy in 3 Gy fractions over 2 weeks) and vorinostat in study participants with histologically-confirmed intrapelvic gastrointestinal carcinoma. Sixteen participants were enrolled into cohorts of escalating vorinostat dose (100 mg, 200 mg, 300 mg, and 400 mg daily). The most common adverse events were grade 1 and 2, among which fatigue and gastrointestinal events were most common. Grade 3 adverse events included fatigue (n = 5), hyponatremia (n = 1), hypokalemia (n = 1), and acneiform rash (n = 1). Of these, treatment related grade 3 events [ie, dose limiting toxicities (DLT)] were observed in 1 of 6 participants at vorinostat 300 mg daily (fatigue and anorexia), and in 2 of 6 participants at the 400 mg daily dose. As a result, the maximum tolerated dose of vorinostat in combination with palliative radiotherapy was determined to be 300mg daily. The study concluded that vorinostat can be safely combined with short term palliative radiotherapy. It should be noted that the adverse events observed in the combination trial overlap with the toxicity profile of vorinostat listed in the package insert.

Anecdotal experience in a patient who was failing standard course of TSEBT is relevant and is described here. This patient's skin lesions were progressing towards the latter half of his TSEBT course, thus, vorinostat was initiated and overlapped with TSEBT in the last 2 weeks. The patient tolerated the combination well without any worsening skin reactions and his skin lesions cleared completely. At one year follow-up, his skin is still in complete remission. Another patient received a combination of romidepsin, another (HDAC) inhibitor, and low-dose (12 Gy) TSEBT. He had CR after the addition of TSEBT, while his skin lesions were stable on romidepsin alone.

Based on preclinical, early clinical data and anecdotal experience, it is anticipated that vorinostat in combination with TSEBT can be administered safely and will be tolerated in participants with MF. In addition, within the recognized limits of a phase 1-2 clinical trial, this study may provide an assessment of the anti-tumor activity of vorinostat in combination with TSEBT in participants with MF and thus allow us to evaluate the radiation-enhancing potential of vorinostat.

This study is a multicenter phase 1-2, randomized, 2-arm trail exploring the efficacy of TSEBT 12 Gy alone vs TSEBT 12 Gy + vorinostat. 12 Gy was selected for this study because it is effective as a rapid debulking agent (with overall response rates of near 100% in the retrospective study and ongoing clinical trial) and can be administered conveniently over 3 weeks. Because of the diminished clinical CR rates associated with TSEBT doses < 30 Gy, it is proposed that combining TSEBT 12 Gy with vorinostat will lead to significantly higher complete response (CR) rates, longer time-to-progression (TTP), and improved quality of life as compared to TSEBT 12 Gy alone. Based on the retrospective study and preliminary experience in the ongoing 12 Gy TSEBT trial, it is hypothesized that 12 Gy is an adequate dose to achieve clinically meaningful outcomes and that the vorinostat may enhance its clinical efficacy while minimizing radiation-associated toxicities due to the shortened treatment duration.

Participants are stratified by MF stage as follows.

* Stage IB: ~10 % skin involvement, with up to 1000/mm3 clone+ Sezary cells in blood.
* Stage IIA: Up to 10 % skin involvement, with up to 1000/mm3 clone+ Sezary cells in blood and clinically abnormal peripheral lymph nodes.
* Stage IIB: One or more tumors 1 cm in diameter, with up to 1000/mm3 clone+ Sezary cells in blood and clinically abnormal peripheral lymph nodes.
* Stage IIIB: Skin erythema >80 % body surface area, with up to 1000/mm3 clone+ Sezary cells in blood and clinically abnormal peripheral lymph nodes.

For detailed staging information, see References: Olsen E, et al. Blood. 2007;110:1713-1722. PMID: 17540844

ELIGIBILITY:
INCLUSION CRITERIA

* Biopsy-confirmed mycosis fungoides (MF); clinical stage IB; IIA; IIB; or IIIB.
* Patients must have failed or have been intolerant to at least one prior systemic or skin-directed therapy. This may include topical steroids if used as primary therapy for MF.
* 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) of ≤ 2.
* White blood cell (WBC) > 2000/uL
* Platelet count > 75,000/mm3
* Absolute neutrophil count (ANC) > 1000.
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x UNL
* Alanine aminotransferase (ALT) ≤ 2.5 x UNL
* Alkaline phosphatase (liver fraction) ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x UNL OR creatinine clearance ≤ 60 mL/min for patients with creatinine levels > 1.5 x institutional ULN
* Potassium level between 3.5 and 4.5
* Magnesium level between 1.5 and 2.5
* Required washout period for prior therapies

  * Topical therapy: 2 weeks
  * Systemic biologic, monoclonal antibody, or chemotherapy: 4 weeks
  * Phototherapy or radiotherapy (excluding TSEBT): 4 weeks
  * Other investigational therapy: 4 weeks
  * Note: patients with rapidly progressive disease may be treated earlier than required washout period; however, such circumstance must be discussed and approved by the protocol director at the primary site (Stanford).
* Women of child-bearing potential (WOCBP) must have negative serum pregnancy test.
* WOCBP must agree to use effective contraception, defined as oral contraceptives, intrauterine devices, double barrier method (condom plus spermicide or diaphragm) or abstain from sexual intercourse. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for 12 consecutive months).
* Male subjects must be willing to use an appropriate method of contraception (eg, condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception (eg, birth control pills) during the study.
* Ability to understand and sign a written informed consent document.
* Ability to comply with the treatment schedule

EXCLUSION CRITERIA

* Prior courses of TSEBT (Note : localized skin-directed radiotherapy is allowed if administered at least 4 weeks prior to initiation on study).
* Concomitant use of any anti-cancer therapy or immune modifier.
* Receiving colony stimulating factors.
* Prior allogeneic or autologous transplant.
* Active infection or have received intravenous antibiotics, antiviral, or antifungal agents within 2 weeks prior to the start of the study drug.
* Known history of human immunodeficiency virus (HIV), hepatitis B or C.
* History of prior malignancy with the exception of cervical intraepithelial neoplasia, non-melanoma skin cancer, and adequately treated localized prostate carcinoma (PSA < 1.0). Patients with a history of other malignancies must have undergone potentially curative therapy and have no evidence of that disease for 5 years.
* Uncontrolled intercurrent illness, condition, or circumstances that could limit compliance with the study, including, but not limited to the following: active infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, unstable angina pectoris, medically significant cardiac arrhythmia, uncontrolled diabetes mellitus or hypertension, or psychiatric conditions.
* Medically significant cardiac event in prior 6 months (ie, myocardial infarction, cardiac surgery.
* Congenital long QT syndrome.
* QTc interval > 480 msec on screening ECG.
* Proven or suspected stage IV disease including patients with B2 (Sezary syndrome); N3 (frank LN disease); or M1 (visceral disease) categories; presence of reactive or dermatopathic lymphadenopathy (N1-2) or limited blood involvement (B1) is permitted.
* Pregnant or lactating.
* Unwilling to use reliable birth control methods.
* Any other medical issue, including laboratory abnormalities, deemed by the Investigator to be likely to interfere with patient participation.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Kim, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zelenetz AD, Abramson JS, Advani RH, Andreadis CB, Byrd JC, Czuczman MS, Fayad L, Forero A, Glenn MJ, Gockerman JP, Gordon LI, Harris NL, Hoppe RT, Horwitz SM, Kaminski MS, Kim YH, Lacasce AS, Mughal TI, Nademanee A, Porcu P, Press O, Prosnitz L, Reddy N, Smith MR, Sokol L, Swinnen L, Vose JM, Wierda WG, Yahalom J, Yunus F. NCCN Clinical Practice Guidelines in Oncology: non-Hodgkin's lymphomas. J Natl Compr Canc Netw. 2010 Mar;8(3):288-334. doi: 10.6004/jnccn.2010.0021. No abstract available. PMID 20202462
- [Background] Olsen E, Vonderheid E, Pimpinelli N, Willemze R, Kim Y, Knobler R, Zackheim H, Duvic M, Estrach T, Lamberg S, Wood G, Dummer R, Ranki A, Burg G, Heald P, Pittelkow M, Bernengo MG, Sterry W, Laroche L, Trautinger F, Whittaker S; ISCL/EORTC. Revisions to the staging and classification of mycosis fungoides and Sezary syndrome: a proposal of the International Society for Cutaneous Lymphomas (ISCL) and the cutaneous lymphoma task force of the European Organization of Research and Treatment of Cancer (EORTC). Blood. 2007 Sep 15;110(6):1713-22. doi: 10.1182/blood-2007-03-055749. Epub 2007 May 31. PMID 17540844

RESULTS

PARTICIPANT FLOW:
Groups:
- TSEBT Only: • TSEBT as 12 grey (Gy), fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment); 4 days each week; for a total of 3 weeks.
- TSEBT Plus Vorinostat: * TSEBT as 12 grey (Gy), fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment); 4 days each week; for a total of 3 weeks.
  * Vorinostat 400 mg/day continuing for 8 weeks total.
Period: Overall Study
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Patient started non-protocol therapy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TSEBT Plus Vorinostat: * TSEBT as 12 grey (Gy), fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment); 4 days each week; for a total of 3 weeks.
  * Vorinostat 400 mg/day concurrent and continuing for 8 weeks total.
- Total: Total of all reporting groups
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Clinical Stage [Count of Participants; unit: Participants] — Participants are stratified by MF stage as follows.
  * Stage IB: ~10 % skin involvement, with up to 1000/mm3 clone+ Sezary cells in blood. No abnormal lymph nodes.
  * Stage IIA: Up to 10% skin involvement, with up to 1000/mm3 clone+ Sezary cells in blood & clinically abnormal peripheral lymph nodes.
  * Stage IIB: One or more tumors 1 cm in diameter, with up to 1000/mm3 clone+ Sezary cells in blood & clinically abnormal peripheral lymph nodes.
  * Stage IIIB: Skin erythema >80 % body surface area, with up to 1000/mm3 clone+ Sezary cells in blood & clinically abnormal peripheral lymph nodes.
  Participants
    Mycosis fungoides, Stage IB | 9 | 8 | 17
    Mycosis fungoides, Stage IIA | 2 | 2 | 4
    Mycosis fungoides, Stage IIB | 2 | 3 | 5
    Mycosis fungoides, Stage IIIB | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical Response (CCR)
Description: Complete Clinical Response (CCR) at week 8 as determined by an Modified Severity-Weighted Assessment Tool (mSWAT) score of 0. mSWAT is an objective, quantitative, severity-weighted method to assess the extent of mycosis fungoides (MF) lesions, and is determined by total body surface area (%TBSA) of the lesion by a severity-weighting factor (1 = patch; 2 = plaque; 4 = tumor). O% TBSA produces a product of 0, indicating complete response.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Number analyzed (Participants) | 14 | 13
Participants | 3 | 3

2. Secondary Outcome: Safety and Tolerability as Measured by Severity and Frequency of Adverse Events
Description: Adverse events occurring at least 10% out of evaluable participants, and it's corresponding rate in the opposing arm.
Time Frame: Adverse events were collected through 30 days after the last day of study therapy, or until the patient received an non-study treatment for lymphoma, whichever occurred first.
Measure: Number; unit: Number of patients
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Number analyzed (Participants) | 14 | 13
Number of patients
  Alopecia | 7 | 10
  Fatigue | 4 | 10
  Extremity Pain | 9 | 6
  Nausea | 0 | 8
  Dysgeusia | 0 | 4
  Nail Changes | 4 | 1
  Diarrhea | 0 | 3
  Ocular Irritation | 0 | 3
  Radiation Dermatitis | 1 | 3
  Thrombocytopenia | 0 | 3
  Anorexia | 0 | 2
  Dizziness | 0 | 2
  Lymphopenia | 0 | 2
  Pedal Edema | 2 | 1
  Skin Pain | 1 | 2
  Vomiting | 0 | 2
  Xerosis/Dry Skin | 1 | 2

3. Secondary Outcome: Clinical Response Rate (CRR)
Description: Clinical Response Rate (CRR) at week 8 as determined by an Modified Severity-Weighted Assessment Tool (mSWAT) score of 0, consisting of complete response (CR) rate; partial response (PR) rate; stable disease (SD) rate; or progressive disease (PD) rate.
  CR = 100% clearance of skin disease (mSWAT score = 0) PR = 50%to <100% clearance of skin disease as measured by > 50% decrease of mSWAT score compared with baseline SD = Not CR, PR, or PD
  PD = Whichever is met first of:
  1. > 25% increase in skin disease from baseline as measured by > 25% increase of mSWAT score compared with baseline
  2. New tumor (T3) lesions in patients without prior T3 lesions (T1, T2, T4) or
  3. In responders (confirmed), increase in skin disease over nadir by 50% of baseline as measured by mSWAT score of > [nadir + > 50% of baseline]
  4. Relapse applies to any new disease after confirmed CR
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Number analyzed (Participants) | 14 | 13
Participants
  Complete Response (CR) | 3 | 3
  Partial Response | 8 | 10
  Stable Disease | 3 | 0
  Progressive Disease | 0 | 0

4. Secondary Outcome: Duration of Clinical Benefit (Per Protocol Follow-up)
Description: Duration of clinical benefit represents the period of time that clinical response was maintained. Duration of clinical benefit is reported as the median period of time from the initiation of treatment until progressive disease, as measured by the mSWAT skin assessment, and censored at the final per-protocol assessment (48 weeks)
Time Frame: 48 weeks after completion of treatment
Population: The data are reported for the per-protocol period of follow-up (48 weeks).
Measure: Median (Full Range); unit: Weeks
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Number analyzed (Participants) | 14 | 13
Weeks | 48 [9.6 to 48] | 28 [5.7 to 48]

5. Secondary Outcome: Duration of Clinical Benefit (Supplemental Follow-up)
Description: Duration of clinical benefit represents the period of time that clinical response was maintained. Duration of clinical benefit is reported as the median period of time from the initiation of treatment or until progressive disease, as measured by the mSWAT skin assessment.
Time Frame: 140 weeks
Population: The data are reported for the full period for which participant data are available.
Measure: Median (Full Range); unit: weeks
Arm/Group | TSEBT Only | TSEBT Plus Vorinostat
Number analyzed (Participants) | 14 | 13
weeks | 125 [9.6 to 135.1] | 28 [5.7 to 82.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 30 days after the last day of study therapy, or until the patient received an non-study treatment for lymphoma, whichever occurred first.
Groups:
- TSEBT Only: TSEBT (12Gy) per institutional guidelines.
- TSEBT & Vorinostat: TSEBT (12Gy) per institutional guidelines.
  Vorinostat 400 mg daily starting one day prior to the initiation of TSEBT.
Arm/Group | TSEBT Only | TSEBT & Vorinostat
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSEBT Only (N=14) | TSEBT & Vorinostat (N=14)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TSEBT Only (N=14) | TSEBT & Vorinostat (N=14)
Abscess of Head and Neck (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 10
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Psychiatric disorders) | 0 | 2
Blistering of Feet (Skin and subcutaneous tissue disorders) | 1 | 1
Blistering of Lip (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (General disorders) | 0 | 1
Diarrhea (General disorders) | 0 | 3
Dizziness (General disorders) | 0 | 2
Dry Mouth (General disorders) | 0 | 1
Dysgeusia (General disorders) | 0 | 4
Dyspepsia (General disorders) | 0 | 1
Elevated Bilirubin (Blood and lymphatic system disorders) | 0 | 1
Elevated Creatinine (Blood and lymphatic system disorders) | 0 | 1
Extremity Pain (General disorders) | 9 | 10
Eye Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 10
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1 | 1
Hyponatremia (Blood and lymphatic system disorders) | 0 | 1
Jaw Pain (General disorders) | 0 | 1
Leucopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Nail Changes (General disorders) | 4 | 1
Nausea (General disorders) | 0 | 8
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Ocular Irritation (Eye disorders) | 0 | 3
Oral Pain (Lips/Cheilitis) (General disorders) | 1 | 0
Oral Ulcer (General disorders) | 1 | 0
Pedal Edema (General disorders) | 2 | 1
Peeling of Skin on Limbs (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3
Skin Infection (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Pain (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vomiting (General disorders) | 0 | 2
Xerosis/Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Gynecomastia (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No